CLINICAL TRIAL: NCT05099978
Title: Asian Multicenter Prospective Study of Circulating Tumor DNA Sequencing: A-TRAIN
Brief Title: Asian Multicenter Prospective Study of ctDNA Sequencing
Acronym: A-TRAIN
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Cancer Center, Japan (Other Government)
Responsible Party: Sponsor
Other Study IDs: NCCH1905
Record Dates: First submitted 2021-09-21; First posted 2021-10-29 (Actual); Last update posted 2024-09-04 (Actual); Status verified 2023-10

CONDITIONS: Cervical Cancer; Ovarian Clear Cell Carcinoma; Nasopharyngeal Carcinoma; Ovarian Cancer; Endometrial Cancer; Triple Negative Breast Cancer
Keywords: ctDNA; Solid tumor in Asia
MeSH Terms: conditions — Uterine Cervical Neoplasms; Nasopharyngeal Carcinoma; Ovarian Neoplasms; Endometrial Neoplasms; Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Peripheral blood sample and unstained 5-micron formalin-fixed paraffin-embedded (FFPE) tumor tissue section
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- NGS analysis of ctDNA: This study consists of 6 cohorts; cervical cancer(n=100), ovarian clear cell cancer(n=50), nasopharyngeal cancer(n=96), ovarian cancer(n=100), breast cancer(n=100), endometrial cancer(n=60).
  In each cohort, the blood samples will be collected within 2weeks after registration. ctDNA will be extracted from blood samples and somatic gene abnormalities will be analyzed using NGS, PCR, and Sanger sequencing. In addition, the analysis of DNA methylation and RNA sequencing may be performed to obtain information related to gene expression.
  Interventions: Genetic: NGS analysis of ctDNA

INTERVENTIONS:
Genetic: NGS analysis of ctDNA — Diagnostic Test: plasma circulating tumor DNA

SUMMARY:
This study is a genetic analysis of aberrations in circulating tumor DNA (ctDNA) in patients in Asian countries. This study protocol is divided into parts describing several subanalyses that differ in terms of cancer types, analytical methods, participating countries, and participating institutions.

DETAILED DESCRIPTION:
NGS analysis will be performed on cfDNA extracted from peripheral blood samples of target patients to determine the types and incidences of genetic abnormalities. Patient information and gene abnormality data will be integrated, and the types and incidences of gene abnormalities by cancer type will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or older at registration.
2. Diagnosis of cancer which is targeted by each cohort.
3. Metastatic and/or recurrent disease.

Exclusion Criteria:

1. Any other malignancy within 3 years prior to registration, except for adequately treated basal cell or squamous cell skin cancer, or carcinoma in situ of the esophagus, stomach, colon, or cervix.
2. Ongoing chemotherapy. (Chemotherapy-naïve patients or awaiting initiation of the next line of chemotherapy are eligible. There is no limit on the number of prior chemotherapies or on the time from completion of chemotherapy to registration).
3. Ongoing radiation therapy. (There are no limits on the time from completion of radiation therapy to registration).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with metastatic and/or recurrent solid cancer which is targeted by each cohort in Asia.
Sampling Method: Probability Sample
Enrollment: 506 (Estimated)
Dates: Start 2021-11-01 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients with one or more genetic abnormalities among all examination cases | Through study completion, an average of 1 year
  DNA may be extracted from blood or tumor tissue samples, and germline gene abnormality may be analyzed using techniques such as PCR, NGS, and Sanger sequencing.
Percentage of patients with each genetic abnormality among all examination cases | Through study completion, an average of 1 year
  DNA may be extracted from blood or tumor tissue samples, and germline gene abnormality may be analyzed using techniques such as PCR, NGS, and Sanger sequencing.

SECONDARY OUTCOMES:
Genomic abnormalities of ctDNA and tumor tissue will be combined to report the concordance rate | Through study completion, an average of 1 year
  Concordance rate is defined by the sum of concordance on positives with the denominator as the total number of genes in which a genomic alteration is detected, i.e., genes in which alterations are not detected by one of assays are excluded from both the numerator and denominator.

CONTACTS AND LOCATIONS:
Overall Officials: Kan Yonemori, MD, PhD, Principal Investigator — Department of Medical Oncology, National Cancer Cancer Hospital
Locations (19):
- National Cancer Center Hospital, Tokyo, Japan
- Malaysia (4):
  - Sarawak General Hospital, Kuching, Sarawak
  - University Malaya Medicine Centre, Kuala Lumpur, Selangor
  - Hospital Kuala Lumpur, Kuala Lumpur
  - Institut Kanser Negara, Putrajaya
- St. Luke's Medical Center, Manila, Philippines
- Singapore (2):
  - National Cancer Centre of Singapore, Bukit Merah
  - National University Hopital, Kent Ridge
- Severance Hospital, Yonsei University Health System, Seoul, South Korea
- National Taiwan University Hospital, Taipei, Zhongzheng Dist, Taiwan
- Thailand (7):
  - Vajira Hospital, Bangkok
  - Chulalongkorn University, Bangkok
  - Faculty of Medicine Ramathibodi Hospital, Mahidol University, Bangkok
  - Phramongkutklao Hospital, Bangkok
  - Mahidol University by Faculty of Medicine, Siriraj Hospital, Bangkok
  - Chiang Mai University, Chiang Mai
  - Songklanagarind Hospital, Songkhla
- Vietnam (2):
  - K Hospital, Hanoi
  - Ho Chi Minh City Oncology Hospital, Ho Chi Minh City